CLINICAL TRIAL: NCT01926769
Title: A Phase II Study to Determine the Safety and Efficacy of Second-line Treatment With Metformin and Chemotherapy (FOLFOX6 or FOFIRI) in the Second Line Threatment of Advanced Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual rate
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hee Kyung Ahn, Assistant Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-GIRBA-2675
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Previously Treated Advanced Colorectal Cancer
Keywords: Colorectal cancer; Metformin; FOLFOX6; FOFIRI; 5FU; irinotecan; oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Metformin

ARMS (1):
- FOLFOX6+Metformin/FOFIRI+Metformin (Experimental)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
To determine the safety and efficacy of second-line treatment with Metformin and Chemotherapy (FOLFOX6 or FOFIRI) in the second line treatment of advanced colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* histologically confirmted advanced colorectal cancer
* ECOG PS 0-2
* expected life span more than 3months
* normal bone marrow, liver, renal function

Exclusion Criteria:

* 5-FU, oxaliplatin, irinotecan or Metformin Allergic history
* Lactic acidosis, metabolic acidosis
* active infection or severe neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate | one year

SECONDARY OUTCOMES:
Response Rate | one year
Overall Survival | one year
Number of participants with adverse events | one year
Progression Free Survival | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea